CLINICAL TRIAL: NCT02249741
Title: PROSPECTIVE STUDY OF PROFILE OF HEPATIC OSTEODYSTROPHY IN PATIENTS WITH NON-CHOLEASTATIC LIVER CIRRHOSIS AND IMPACT OF BISPHOSPHONATE SUPPLEMENTATION
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dr. Ashish Kumar (Other)
Responsible Party: Sponsor-Investigator, Dr. Ashish Kumar, Associate Professor, Sir Ganga Ram Hospital
Organization: Sir Ganga Ram Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Gastro-2012-RB-1
Record Dates: First submitted 2014-09-23; First posted 2014-09-26 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-09

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis | interventions — Therapeutics; Ibandronic Acid

ARMS (1):
- Patients with osteoporosis (Experimental): Treated with Ibandronic acid as per protocol
  Interventions: Drug: Treated with Ibandronic acid as per protocol

INTERVENTIONS:
Drug: Treated with Ibandronic acid as per protocol — treated with Ibandronic acid at a dose of 150 mg once a month for six months

SUMMARY:
Background and Objectives: Patients with liver cirrhosis are more prone to develop reduced bone mineral density i.e. hepatic osteodystrophy (HOD). It includes both osteopenia and osteoporosis and may lead to increased fracture risks. There is scanty data on prevalence of HOD in Indian population and its treatment outcome. The investigators aimed to determine prevalence of HOD, factors associated with it and the impact of bisphosphonates on bone mineral density in patients with liver cirrhosis.

Patients and Methods: Consecutive patients with liver cirrhosis admitted at Sir Ganga Ram Hospital, New Delhi between August 2012 and July 2013 were enrolled. Patients with chronic kidney disease, hyperparathyroidism and those on steroids were excluded. Bone mineral density (BMD) was measured by dual-energy X-ray absorptiometry (DEXA) at the lumbar spine and femoral neck. Osteopenia and osteoporosis were defined according to WHO criteria. All patients also underwent 25-hydroxy-vitamin-D, sex hormone (testosterone in male and LH and Estradiol in female) and parathyroid hormone (PTH) along with routine investigations. Transient elastography was also done in all patients. Ibandronic acid 150 mg per day orally for six months was given in patients with osteoporosis and DEXA scan repeated.

ELIGIBILITY:
Inclusion Criteria:

1. Liver Cirrhosis
2. Age 18-70 years
3. Informed and written consent

Exclusion Criteria:

1. Chronic renal failure
2. Prolonged steroid use more than 3 months
3. Patients on immunosuppressive therapy
4. Primary hyperparathyroidism
5. Post menopausal women
6. Pregnancy
7. Cushing's syndrome
8. Malignancy
9. HIV Co-infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2012-08; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Improvement in Bone Mineral Density on DEXA scan | 6 months

SECONDARY OUTCOMES:
Incidence of new fractures | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroenterology & Hepatology, Sir Ganga Ram Hospital, New Delhi, New Delhi, India